CLINICAL TRIAL: NCT03283358
Title: Person-centered Follow up and Health Promotion Program After Revascularization for Intermittent Claudication
Acronym: FASTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anneli Linné, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FASTIC-1
Record Dates: First submitted 2016-06-13; First posted 2017-09-14 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Intermittent Claudication
Keywords: Prevention and control
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Person-centered follow up (Experimental): The intervention program is a person-centered health promotion program led by a nurse and consists of two telephone calls (15 minutes each) at two weeks and nine months after surgical treatment for Intermittent Claudication and three visits (45 - 60 min) at six weeks, six months and one year after treatment. The program includes a baseline assessment, an individual plan for self-care and educational information about Intermittent Claudication, received treatment and secondary prevention (medication and modifiable risk factors). The purpose is to enhance self-care in terms of adherence to medication and to recommended changes of lifestyle.
  Interventions: Behavioral: Person-centered follow up
- Standard follow up (No Intervention): Standard follow-up consist of two follow up appointments á 20 minutes at four-six weeks and one year after surgical treatment of Intermittent Claudication. The patients meet a vascular surgeon at the first follow up and a vascular nurse or a surgeon at the second follow up visit.

INTERVENTIONS:
Behavioral: Person-centered follow up
  Arms: Person-centered follow up

SUMMARY:
The overall aim of the study is to evaluate a nurse-led intervention (person-centered follow up and health promotion) program in comparison to standard follow up for patients treated with surgical or endovascular revascularization of Intermittent Claudication.

DETAILED DESCRIPTION:
Specific Aims:

1. To evaluate the effect of the intervention program on patient's adherence to medication (anticoagulant agents, antiplatelet agents and lipid-lowering agents), risk modification and surgical treatment outcomes
2. To investigate the effect of the intervention program on patient reported outcomes
3. To investigate the effect of the intervention program on patient reported experiences
4. To investigate the long-term effect of the intervention program on mortality, cause of death, occurrence/recurrence of cardiovascular disease up to 10 years after the surgical/endovascular treatment
5. To compare patient-reported adherence to medication and patient data registry adherence to medication

Hypothesis: Participants in the Intervention Group have better adherence to prescribed medication and a reduced risk for 10-year predicted coronary heart disease (CHD) compared to participants in the Control Group.

Study population:

Patients with Intermittent Claudication scheduled for revascularization, through open surgery or endovascular method, in Stockholm will be screened for inclusion. After informed consent, the participants will be randomized to either Intervention Group or Control Group. Those participants who couldn't receive revascularization after giving consent will be withdrawn from the study and counted as drop outs. Power analysis has showed a required sample size of 186 participants to detect a statistically significant increase in adherence to medication from 50% to 70% (power 0.80, significance value 0.05, two-sided). Expecting 10% drop-out we plan to recruit 210 participants.

Data collection:

Data on primary and secondary outcomes, serum cholesterol, smoking status, serum carbon monoxide, Hba1c, BMI, waist circumference, physical exercise, diet, alcohol consumption, graft patency, re-intervention, hospitalization during the study year, mortality and patient characteristics/demographics will be collected at baseline and one year after treatment. All data will be registered at a local research data base at Karolinska Institutet. All patient-reported outcomes will be collected using web-based questionnaires linked to the data base.

Data analysis:

Comparisons between the Intervention Group and the Control Group will be made using t-test and ANOVA for repeated-measures or Wilcoxon rank-signed test and Kruskall-Wallis according to the underlying distribution for continuous data, and Fischers Exact test for categorical data. Logistic regression analysis will also be performed to adjust for confounding factors. All analyses will be performed according to the Intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who is scheduled for revascularization, through open and/or endovascular surgery for IC diagnosed according to Diagnosis Related Group (DRG) with I70.2 or I739B

Exclusion Criteria:

* Patients not treated through surgery or revascularization
* Patients diagnosed with dementia
* Patients discharge to a nursery home,
* Patients not accountable for administrating their own medications
* Patients with a survival expectancy less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Adherence to medication | One year after surgical or endovascular treatment for Intermittent Claudication
  Adherence to medication (anticoagulant agents, antiplatelet agents and lipid-lowering agents) according to the Swedish Prescribed Drug Registry (PDR). dispensed anticoagulant agents, antiplatelet agents (ATC-register B01A) and lipid-lowering agents (ATC-register C10). Those participants who have fetched both medications for the second refill after treatment will be considered adherent.

SECONDARY OUTCOMES:
Risk for 10-year predicted coronary heart disease (CHD) | One year after surgical or endovascular treatment for Intermittent Claudication
  Changes in risk for CHD within 10-years measured by Framingham Risk Score (FRHS).

OTHER OUTCOMES:
Patient reported adherence to medication | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported adherence to medication (anticoagulant agents, antiplatelet agents and lipid-lowering agents).
Generic Health-related Quality of Life (HRQOL) | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported generic HrQoL measured by EQ-5D
Condition specific Health-related Quality of Life (HRQOL) | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported specific HrQoL measured by VascQol-6
Beliefs on medication | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported beliefs on medication measured by Beliefs about Meicines Questionnaire (BMQ)
Self-efficacy | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported Self-efficacy measured by Swedish Version of the General Self-Efficacy Scale
Health literacy | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-reported health literacy measured by HLS-EU-Q16 SE
Patient-experienced quality of care | One year after surgical or endovascular treatment for Intermittent Claudication
  Patient-experienced quality of care measured by Quality of Care from Patient's Perspective (Swedish version of QPP)
Mortality | Ten years after surgical or endovascular treatment for Intermittent Claudication
  Data on mortality will be extracted from the National Patient Registry and Stockholm County Council's administrative data (VårdanalysdataLager - VAL).
Cardiovascular disease | Ten years after surgical or endovascular treatment for Intermittent Claudication
  Data on occurrence/reoccurrence of cardiovascular disease with hospitalization will be extracted from the National Patient Registry and Stockholm County Council's administrative data (VårdanalysdataLager - VAL).

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Linné, MD, PhD, Principal Investigator — Karolinska Institutet, Department of Clinical Science and Education, Södersjukhuset
Locations (2):
- Sweden (2):
  - Department of Surgery, Unit of Vascular Surgery, Södersjukhuset, Stockholm
  - Karolinska University Hospital, Dept of Vascular Surgery, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haile ST, Olsson M, Lindstrand R, Loof H, Linne A, Johansson UB, Joelsson-Alm E. Patient Reported Experiences of Receiving Person-Centred, Nurse-Led Follow-Up After Revascularisation for Intermittent Claudication: Secondary Analysis of a Randomised Controlled Trial. J Clin Nurs. 2025 Jul;34(7):3003-3016. doi: 10.1111/jocn.17762. Epub 2025 May 20. PMID 40390575
- [Derived] Haile S, Linne A, Johansson UB, Joelsson-Alm E. Follow-up after surgical treatment for intermittent claudication (FASTIC): a study protocol for a multicentre randomised controlled clinical trial. BMC Nurs. 2020 Jun 4;19:45. doi: 10.1186/s12912-020-00437-7. eCollection 2020. PMID 32518518